CLINICAL TRIAL: NCT01062555
Title: Calcineurin-Sparing in a Steroid-free Maintenance Immunosuppression Protocol After Kidney Transplantation
Brief Title: Calcineurin Inhibitor Sparing After Kidney Transplantation
Acronym: CNI-Sparing
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Roche Pharma AG (Industry); Wyeth is now a wholly owned subsidiary of Pfizer (Industry); Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0604M85327
Record Dates: First submitted 2010-02-03; First posted 2010-02-04 (Estimated); Results first posted 2020-12-14 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-11

CONDITIONS: CNI Side Effects
MeSH Terms: interventions — Cyclosporine; Mycophenolic Acid; Cyclosporins; Tacrolimus; cni protein, Drosophila; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Phase I Arm 1 (Active Comparator): CSA and MMF
  Interventions: Drug: Cyclosporine & Cellcept
- Phase I Arm 2 (Active Comparator): FK and MMF
  Interventions: Drug: Prograf & Cellcept
- Phase II Arm 1 (Active Comparator): Low CNI and MMF
  Interventions: Drug: Low Dose CNI (Cyclosporine or FK) and Cellcept
- Phase II Arm 2 (Active Comparator): Rapa and MMF
  Interventions: Drug: Rapamune and Cellcept

INTERVENTIONS:
Drug: Cyclosporine & Cellcept — Dose and frequency determined as usual by transplant physicians. The drugs are not experimental drugs. The study is looking at reducing negative side effects of some of the drugs.
  Other Names: CSA, Gengraf, Neoral, Sandimmune, MMF, Mycophenolate Mofetil
  Arms: Phase I Arm 1
Drug: Prograf & Cellcept — Dose and frequency determined as usual by transplant physicians. The drugs are not experimental drugs. The study is looking at reducing negative side effects of some of the drugs.
  Other Names: FK, Tacrolimus, MMF, Mycophenolate Mofetil
  Arms: Phase I Arm 2
Drug: Low Dose CNI (Cyclosporine or FK) and Cellcept — Dose and frequency determined as usual by transplant physicians. The drugs are not experimental drugs. The study is looking at reducing negative side effects of some of the drugs.
  Other Names: Gengraf, Neoral, Sandimmune, Tacrolimus, Prograf, MMF
  Arms: Phase II Arm 1
Drug: Rapamune and Cellcept — Dose and frequency determined as usual by transplant physicians. The drugs are not experimental drugs. The study is looking at reducing negative side effects of some of the drugs.
  Other Names: Sirolimus, MMF, Mycophenolate Mofetil
  Arms: Phase II Arm 2

SUMMARY:
Reducing drug side effects is a key issue in transplantation. One class of drugs commonly used, calcineurin inhibitors (CNIs), is associated with negative side effects, namely, toxicity to the transplanted kidney. In some patients, this toxicity is thought to be associated with loss of transplant function in those who have had their transplants for many years. The introduction of new immunosuppression medications however, has provided the opportunity to minimize or avoid CNIs, which may reduce the occurrence of toxicity to the kidney.

DETAILED DESCRIPTION:
It is clear that minimizing the use of CNIs may be beneficial to some or all kidney transplant recipients. The purpose of this study is to determine whether minimization of these CNI drugs will improve patient survival rates and long-term kidney function.

If the subject agrees to participate in this research project, they will be randomly assigned to one of two different immunosuppression drug combinations. All of the drugs used in this study are standard FDA Approved immunosuppressive drugs currently in use by transplant patients. It is unclear however, which combination provides a better long-term outcome.

If after six months of being on the study the subject has not experienced a rejection episode that excludes them from participating in the second phase of this study, they will asked whether or not they would like to continue the study. If they decide to participate in Phase II, there will be another randomization to one of two different immunosuppression drug combinations. This will involve either being assigned to a group that will have their CNI dose lowered or a group that will have their CNI drug stopped and replaced with a non-CNI drug called Sirolimus. Phase II begins at 6 months post-transplant and a second consent will be obtained for those who participate in Phase II.

ELIGIBILITY:
Inclusion Criteria:

* Kidney Transplant Recipients > 18 years old
* First or Second Kidney Transplant only

Exclusion Criteria:

* Kidney Transplant Recipients < 18 years old
* Kidney Transplant Recipients who have a history of > 2 kidney transplants
* Kidney Transplant Recipients with an already functioning non-renal transplant
* Kidney Transplant Recipients who receive another organ simultaneously at the same time of their kidney transplant (example: Kidney/pancreas, kidney/liver)
* Non-skin malignancy with 2 years previous to enrollment
* Donor Specific Antibodies to kidney donor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 527 (Actual)
Dates: Start 2006-10-01 (Actual); Primary Completion 2014-04-03 (Actual); Study Completion 2014-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Matas, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All patients consented at time of transplant for phase 1. At 6 months post-transplant, patients were re-consented for phase 2. All patients represented for phase 2 were included for phase 1. Patients who were not re-consented for phase 2, were followed for 7 years under phase 1 protocol.
Period: Phase 1
Arm/Group | Phase I Arm 1 | Phase I Arm 2 | Phase II Arm 1 | Phase II Arm 2
Started | 266 | 261 | 0 | 0
Completed | 243 | 235 | 0 | 0
Not Completed | 23 | 26 | 0 | 0
Not completed — Death | 10 | 17 | 0 | 0
Not completed — Graft Failure | 12 | 8 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0
Period: Phase 2
Arm/Group | Phase I Arm 1 | Phase I Arm 2 | Phase II Arm 1 | Phase II Arm 2
Started | 0 | 0 | 86 | 87
Completed | 0 | 0 | 71 | 53
Not Completed | 0 | 0 | 15 | 34
Not completed — Death | 0 | 0 | 8 | 3
Not completed — Graft failure | 0 | 0 | 7 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 7
Not completed — Protocol Violation | 0 | 0 | 0 | 3
Not completed — Physician Decision | 0 | 0 | 0 | 17

BASELINE CHARACTERISTICS:
Groups:
- Arm1 (Phase 1 & 2): Participants from Phase 1, Arm 1 (CSA and MMF) and participants from Phase 2, Arm 1 (Low CNI and MMF)
- Arm 2 (Phase 1 & 2): Participants from Phase 1, Arm 2 (FK and MMF) and participants from Phase 2, Arm 2 (Rapa and MMF)
- Total: Total of all reporting groups
Arm/Group | Arm1 (Phase 1 & 2) | Arm 2 (Phase 1 & 2) | Total
Number analyzed (Participants) | 266 | 261 | 527
Age, Categorical [Count of Participants; unit: Participants] — Population: This study had a sequential enrollment. Not all of the participants from phase one moved on to phase two, which is why phase two has a smaller number of participants analyzed.
  Participants
    Phase 1: <=18 years | 0 | 1 | 1
    Phase 1: Between 18 and 65 years | 214 | 215 | 429
    Phase 1: >=65 years | 52 | 45 | 97
    Phase 2: number analyzed (Participants) | 86 | 87 | 173
    Phase 2: <=18 years | 0 | 0 | 0
    Phase 2: Between 18 and 65 years | 67 | 74 | 141
    Phase 2: >=65 years | 19 | 13 | 32
Sex: Female, Male [Count of Participants; unit: Participants] — Population: This study had a sequential enrollment. Not all of the participants from phase one moved on to phase two, which is why phase two has a smaller number of participants analyzed.
  Participants
    Phase 1: Female | 89 | 94 | 183
    Phase 1: Male | 177 | 167 | 344
    Phase 2: number analyzed (Participants) | 86 | 87 | 173
    Phase 2: Female | 23 | 31 | 54
    Phase 2: Male | 63 | 56 | 119
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: This study had a sequential enrollment. Not all of the participants from phase one moved on to phase two, which is why phase two has a smaller number of participants analyzed.
  Participants
    Phase 1: American Indian or Alaska Native | 6 | 9 | 15
    Phase 1: Asian | 18 | 13 | 31
    Phase 1: Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
    Phase 1: Black or African American | 19 | 12 | 31
    Phase 1: White | 221 | 227 | 448
    Phase 1: More than one race | 0 | 0 | 0
    Phase 1: Unknown or Not Reported | 0 | 0 | 0
    Phase 2: number analyzed (Participants) | 86 | 87 | 173
    Phase 2: American Indian or Alaska Native | 1 | 4 | 5
    Phase 2: Asian | 2 | 7 | 9
    Phase 2: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Phase 2: Black or African American | 6 | 6 | 12
    Phase 2: White | 77 | 70 | 147
    Phase 2: More than one race | 0 | 0 | 0
    Phase 2: Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 266 | 261 | 527

OUTCOME MEASURES:

1. Primary Outcome: Phase I: The Minimization of Negative Side Effects - Patient Survival
Description: The percentage of patients alive at 6 month post transplant.
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Phase I Arm 1 | Phase I Arm 2
Number analyzed (Participants) | 266 | 261
percentage of participants | 99 | 98

2. Primary Outcome: Phase II: The Minimization of Negative Side Effects - Patient Survival
Description: The percentage of patients alive at 7 years post transplant or at the end of study activities. Not all participants completed 7-year follow-up.
Time Frame: up to 7 years
Measure: Number; unit: percentage of participants
Arm/Group | Phase II Arm 1 | Phase II Arm 2
Number analyzed (Participants) | 86 | 87
percentage of participants | 89 | 85

3. Primary Outcome: Phase I: The Minimization of Negative Side Effects - Graft Survival
Description: Percent of participants at 6 months with a functioning graft (without graft failure).
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Phase I Arm 1 | Phase I Arm 2
Number analyzed (Participants) | 266 | 261
percentage of participants | 99 | 99

4. Primary Outcome: Phase II: The Minimization of Negative Side Effects - Graft Survival
Description: The percentage of patients with a functioning graft (without graft failure) at 7 years post transplant or at the end of study activities. Not all participants completed 7-year follow-up.
Time Frame: up to 7 years
Measure: Number; unit: percentage of participants
Arm/Group | Phase II Arm 1 | Phase II Arm 2
Number analyzed (Participants) | 86 | 87
percentage of participants | 80 | 78

5. Primary Outcome: Phase I: Acute Rejection-Free Survival
Description: Percent of participants at 6 months without acute rejection.
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Phase I Arm 1 | Phase I Arm 2
Number analyzed (Participants) | 266 | 261
percentage of participants | 80 | 85

6. Primary Outcome: Phase II: Acute Rejection-Free Survival
Description: The percentage of patients without acute rejection at 7 years post transplant or at the end of study activities. Not all participants completed 7-year follow-up.
Time Frame: up to 7 years
Measure: Number; unit: percentage of participants
Arm/Group | Phase II Arm 1 | Phase II Arm 2
Number analyzed (Participants) | 86 | 87
percentage of participants | 76 | 81

ADVERSE EVENTS:
Time Frame: Phase 1 - 6 months Phase 2 - 7 years
Description: Non-serious adverse events were not collected.
Arm/Group | Phase I Arm 1 | Phase I Arm 2 | Phase II Arm 1 | Phase II Arm 2
All-Cause Mortality (participants affected / at risk) | 10/266 | 17/261 | 8/86 | 3/87
Serious Adverse Events (participants affected / at risk) | 0/266 | 0/261 | 0/86 | 0/87
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes